CLINICAL TRIAL: NCT06680518
Title: Prospective, Randomized Study of Tourniquet Use in Hallux Valgus Surgery
Brief Title: Tourniquet Use in Hallux Valgus Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint Jean, France (Other)
Responsible Party: Principal Investigator, Wayan HEBRARD, Doctor, Clinique Saint Jean, France
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2024-A01589-38
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hallux Valgus
Keywords: hallux valgus; tourniquet
MeSH Terms: conditions — Hallux Valgus | interventions — Tourniquets

STUDY DESIGN:
Intervention Model Description: The patient will be his or her own control, with one foot operated with a tourniquet and the other without.
  Once the patient has been included, the surgeon will open the randomization envelope to determine which foot will receive the tourniquet. He will operate on the left foot first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm with tourniquet (Active Comparator): The surgeon will use the tourniquet as usual.
  Interventions: Other: tourniquet
- Arm without tourniquet (Experimental): The surgeon will operate without the aid of a tourniquet
  Interventions: Other: No tourniquet

INTERVENTIONS:
Other: tourniquet — peroperation tourniquet
  Arms: Arm with tourniquet
Other: No tourniquet — no tourniquet during surgery
  Arms: Arm without tourniquet

SUMMARY:
Prospective, single-center, randomized interventional clinical trial of tourniquet use in hallux valgus surgery. Patients will be their own controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 who has been informed and has signed the consent form
* Patient to be operated on for bilateral hallux valgus with no difference in the procedure performed between the 2 feet, the deformity must not differ by more than 10° (angle M1P1) between the 2 sides.
* Surgery planned on the same day for both feet

Exclusion Criteria:

* Arthritic hallux valgus requiring arthrodesis
* Inflammatory pathology (rheumatoid arthritis, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Average pain in the first week after surgery | first week after surgery
  Comparison between the 2 groups of the average VAS over the first week following surgery, from 0 to 100 points, 0 being the value where the patient has no pain and 100 the maximum pain value.

SECONDARY OUTCOMES:
Edema | Day 10 after surgery
  Measurement of foot edema at D10 during the consultation, taking the difference in cm between the postoperative measurement and the preoperative measurement.
Complications | first week after surgery
  Occurrence of complications specific to tourniquet use as a percentage in each arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique St Jean Sud de France, Saint-Jean-de-Védas, France

IPD SHARING:
Plan to Share IPD: Undecided